CLINICAL TRIAL: NCT03307174
Title: A Prospective, Randomized Analysis of Epidural Anesthesia Using Programmed Intermittent Epidural Boluses Versus Continuous Epidural Infusion in Patients Undergoing Abdominal Surgery.
Brief Title: Programmed Intermittent Bolus Dosing Versus Continuous Epidural Infusion for Epidural Analgesia in Abdominal Surgery.
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 15-18354
Record Dates: First submitted 2017-10-05; First posted 2017-10-11 (Actual); Results first posted 2020-05-12 (Actual); Last update posted 2020-05-12 (Actual); Status verified 2020-04

CONDITIONS: Pain, Acute
MeSH Terms: conditions — Acute Pain | interventions — Bupivacaine; Fentanyl

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Continuous epidural infusion (Active Comparator): At our institution, the most commonly utilized form of administration of medication through an epidural (our active comparator/control) is as follows:
  Combination of 0.0625% bupivacaine with 2mcg/ml of fentanyl infused at a constant rate of 8ml/hr. The patient has the ability to self administer patient controlled epidural analgesia of 2ml of the epidural medication with a lock out period of 15 min. The total maximum volume of epidural medication each hour is 16ml. These settings are managed and controlled by a epidural medication pump.
  Additional oral and intravenous analgesia medications are available as scheduled and pro re nata.
  Interventions: Drug: Bupivacaine; Drug: Fentanyl
- Programmed intermittent epidural bolus (Experimental): For the programmed intermittent epidural bolus group:
  Combination of 0.0625% bupivacaine with 2mcg/ml of fentanyl will be administered as a bolus of 4ml every 30 minutes. The patient has the ability to self administer patient controlled epidural analgesia of 2ml of the epidural medication with a lock out period of 10 min. The total maximum volume of epidural medication each hour is 16ml. These settings are managed and controlled by a epidural medication pump.
  Additional oral and intravenous analgesia medications are available as scheduled and pro re nata.
  Interventions: Drug: Bupivacaine; Drug: Fentanyl

INTERVENTIONS:
Drug: Bupivacaine
  Other Names: 0.0625% bupivacaine
Drug: Fentanyl
  Other Names: 2mcg/ml fentanyl

SUMMARY:
Epidurals are an effective means for providing neuraxial anesthesia and analgesia. Prior studies in labor epidurals have demonstrated that a programmed intermittent bolus application of local anesthesia can improve pain control by reducing the amount of local anesthetic required as well as improve patient satisfaction when compared to continuous epidural infusions. The effects of programmed intermittent bolus of epidural local anesthetics compared to continuous epidural infusions in a surgical setting have yet to be elucidated. Our goal is to evaluate the use of programmed intermittent bolus compared to continuous epidural infusion in a surgical patient population. We plan to enroll patients already undergoing abdominal surgeries including colorectal, gynecologic, surgical oncology, urological where epidural anesthesia can be employed. The primary endpoints of the study will be the total local anesthetic consumption and total opioid consumption as surrogate markers for the quality of epidural anesthesia. Secondary endpoints are pain scores and functional measurements, patient satisfaction, and incidence of hypotension.

DETAILED DESCRIPTION:
See brief summary

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesia physical classification I - III, scheduled for surgery with anticipated an epidural anesthesia (including but not limited to colorectal, surgical oncology, urology, gynecology) as part of their perioperative treatment

Exclusion Criteria:

* Age younger than 18 years of age, non-English speaking, contraindication for neuraxial anesthesia (such as, but not limited to coagulopathy, infection at site, allergy to local anesthetic), preexisting neurologic deficits, inability to consent due to cognitive dysfunction, patients with pain numeric rating score > 5 each day for greater than 3 months, daily opioid consumption > 100 oral morphine equivalents for 14 consecutive days prior to surgery, patient refusal.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2016-04-14 (Actual); Primary Completion 2019-02-28 (Actual); Study Completion 2019-02-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Matthias Behrends, MD, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California San Francisco, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were enrolled between December 2016 to December 2018
Pre-assignment Details: Patients were not randomized to study groups if epidurals were not able to be successfully placed.
  2 subjects in the CEI group were no included in the analysis due to missing data
  1 subject in the PIEB group was not included in the analysis due to missing data
Groups:
- Continuous Epidural Infusion: At our institution, the most commonly utilized form of administration of medication through an epidural (our active comparator/control) is as follows:
  Combination of 0.0625% bupivacaine with 2mcg/ml of fentanyl infused at a constant rate of 8ml/hr. The patient has the ability to self administer patient controlled epidural analgesia of 2ml of the epidural medication with a lock out period of 15 min. The total maximum volume of epidural medication each hour is 16ml. These settings are managed and controlled by a epidural medication pump.
  Additional oral and intravenous analgesia medications are available as scheduled and pro re nata.
  Bupivacaine
  Fentanyl
- Programmed Intermittent Epidural Bolus: For the programmed intermittent epidural bolus group:
  Combination of 0.0625% bupivacaine with 2mcg/ml of fentanyl will be administered as a bolus of 4ml every 30 minutes. The patient has the ability to self administer patient controlled epidural analgesia of 2ml of the epidural medication with a lock out period of 10 min. The total maximum volume of epidural medication each hour is 16ml. These settings are managed and controlled by a epidural medication pump.
  Additional oral and intravenous analgesia medications are available as scheduled and pro re nata.
  Bupivacaine
  Fentanyl
Period: Overall Study
Arm/Group | Continuous Epidural Infusion | Programmed Intermittent Epidural Bolus
Started | 60 | 60
Completed | 46 | 53
Not Completed | 14 | 7
Not completed — Unplanned ICU Administrion | 5 | 3
Not completed — Aborted Surgery | 1 | 2
Not completed — Hypotension | 6 | 0
Not completed — Nonfunctional epidural | 1 | 1
Not completed — Planned epidural removal | 1 | 0
Not completed — Intrathecal catheter placement | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Continuous Epidural Infusion | Programmed Intermittent Epidural Bolus | Total
Number analyzed (Participants) | 60 | 60 | 120
Age, Continuous [Mean (Standard Deviation); unit: years] | 58 (14) | 55 (16) | 57 (15)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 42 | 43 | 85
  Male | 18 | 17 | 35
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 42 | 40 | 82
  Latinx | 7 | 9 | 16
  Black/African American | 0 | 1 | 1
  Asian/Pacific Islander | 11 | 10 | 21
Home Medication Use [Count of Participants; unit: Participants]
  Acetaminophen | 13 | 16 | 29
  NSAIDS | 14 | 11 | 25
  Gabapentinoids | 2 | 4 | 6
  TCA/SNRI | 0 | 0 | 0
Daily opioid consumption [Median (Inter-Quartile Range); unit: MME] | 0 [0 to 0] | 0 [0 to 0] | 0 [0 to 0]
Pain Severity [Median (Inter-Quartile Range); unit: units on a scale] — Minimum of 0, maximum of 10. 10 indicates higher severity of pain.
  units on a scale
    Current Pain | 0 [0 to 0] | 0 [0 to 0] | 0 [0 to 0]
    Worst Pain | 2 [0 to 6] | 4 [0 to 7] | 3 [0 to 7]
    Least Pain | 0 [0 to 1] | 0 [0 to 2] | 0 [0 to 1]
    Average Pain | 1 [0 to 4] | 2 [0 to 4] | 1 [0 to 4]
Average Pain Interference [Median (Inter-Quartile Range); unit: units on a scale] — Minimum of 0, maximum of 10. 10 indicates more severe interference of activities due to pain.
  units on a scale | 1 [0 to 3] | 2 [0 to 6] | 1 [0 to 4]
World Health Organization Disability Assessment Schedule 2.0 [Mean (Inter-Quartile Range); unit: units on a scale] — Minimum of 0, maximum of 100. Score of 100 indicates fully disabled
  units on a scale | 12 [4 to 30] | 19 [12 to 32] | 17 [8 to 31]
HADS Anxiety Score [Count of Participants; unit: Participants]
  None | 35 | 34 | 69
  Mild | 14 | 14 | 28
  Moderate | 7 | 9 | 16
  Severe | 4 | 2 | 6
Depression HADS Score [Count of Participants; unit: Participants]
  None | 50 | 45 | 95
  Mild | 4 | 11 | 15
  Moderate | 5 | 3 | 8
  Severe | 1 | 0 | 1
Length of Epidural Therapy [Median (Inter-Quartile Range); unit: Days] | 2 [1 to 3] | 2 [1 to 3] | 2 [1 to 3]
Type of Surgery [Count of Participants; unit: Participants]
  Upper GI (gastric, small intestine) | 8 | 3 | 11
  Lower GI (colorectal) | 18 | 17 | 35
  Hepatobiliary | 13 | 19 | 32
  Gynecologic | 21 | 21 | 42
Intraoperative Opioids [Median (Inter-Quartile Range); unit: MME] | 38 [18 to 60] | 44 [16 to 61] | 39 [16 to 60]

OUTCOME MEASURES:

1. Primary Outcome: Total Local Anesthetic Utilized in First 24 Hours
Description: Total local anesthetic consumed while epidural in place, recorded on infusion pump
Time Frame: In first 24 hours
Population: Note that 2 patients in the CEI group and 1 patient in the PIEB group was not included in the analysis due to missing data.
Measure: Median (Inter-Quartile Range); unit: mg
Arm/Group | Continuous Epidural Infusion | Programmed Intermittent Epidural Bolus
Number analyzed (Participants) | 44 | 52
mg | 126 [120 to 134] | 123 [115 to 136]
Statistical Analysis 1: Comparison: Continuous Epidural Infusion vs Programmed Intermittent Epidural Bolus; Test type: Superiority; p = 0.74, Wilcoxon (Mann-Whitney)

2. Secondary Outcome: Total Opioid Consumed
Description: Total opioid consumed (intravenous or po) while epidural in place
Time Frame: While epidural in place (up to 72 hours post operatively)
Measure: Median (Inter-Quartile Range); unit: MME
Arm/Group | Continuous Epidural Infusion | Programmed Intermittent Epidural Bolus
Number analyzed (Participants) | 44 | 52
MME
  24 hours postoperatively | 12 [0 to 28] | 16 [0 to 27]
  24 - 48 hours postoperatively | 0 [0 to 25] | 0 [0 to 30]
  48 - 72 hrs postoperatively | 0 [0 to 21] | 1 [0 to 18]

3. Secondary Outcome: Patient Satisfaction Score
Description: Ranked patient satisfaction scores while epidural in place. Measured by modified pain inventory.
  Minimum is 0, maximum of 10. 10 indicates highest patient satisfaction.
Time Frame: While epidural in place (up to 72 hours postoperatively)
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Continuous Epidural Infusion | Programmed Intermittent Epidural Bolus
Number analyzed (Participants) | 44 | 52
score on a scale
  24 hours postoperatively | 9 [8 to 10] | 8 [6.5 to 10]
  24 - 48 hours postoperatively | 9 [7 to 10] | 9 [7.3 to 10]
  48 - 72 hours postoperatively | 9 [7 to 10] | 9 [8 to 10]

4. Secondary Outcome: Average Pain Severity
Description: Measured by modified pain inventory on a daily basis while epidural in place. Minimum is 0, maximum is 10. 10 indicates highest pain severity.
Time Frame: While epidural in place (up to 72 hours postoperatively)
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Continuous Epidural Infusion | Programmed Intermittent Epidural Bolus
Number analyzed (Participants) | 44 | 52
units on a scale
  24 hours postoperatively | 3 [1 to 4] | 5 [2 to 5]
  24 - 48 hours postoperatively | 3 [1 to 4] | 2 [1 to 5]
  48 - 72 hours postoperatively | 3 [1 to 4] | 3 [1 to 4]

5. Secondary Outcome: Incidence of Hypotension
Description: Most common side effect post-operatively with epidural anesthesia. Documented by recorded vitals signs, fluid resuscitation, and temporary cessation of epidural medication.
Time Frame: While epidural in place (24 hours postoperatively)
Measure: Count of Participants; unit: Participants
Arm/Group | Continuous Epidural Infusion | Programmed Intermittent Epidural Bolus
Number analyzed (Participants) | 44 | 52
Participants | 9 | 18

6. Secondary Outcome: Worst Reported 24 Hour Pain
Description: Minimum is 0, maximum is 10. 10 indicates highest pain severity.
Time Frame: While epidural in place (up to 72 hours postoperatively)
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Continuous Epidural Infusion | Programmed Intermittent Epidural Bolus
Number analyzed (Participants) | 44 | 52
score on a scale
  24 hours postoperatively | 5 [2 to 7] | 8 [4 to 9]
  24 - 48 hours postoperatively | 6 [3 to 8] | 6 [3 to 8]
  48 - 72 hours postoperativley | 7 [5 to 8] | 6 [3 to 8]

7. Secondary Outcome: Average Pain Interference
Description: Minimum is 0, maximum is 10. 10 indicates highest pain interference.
Time Frame: While epidural in place (up to 72 hours postoperatively)
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Continuous Epidural Infusion | Programmed Intermittent Epidural Bolus
Number analyzed (Participants) | 44 | 52
score on a scale
  24 hours postoperatively | 2 [0 to 4] | 3 [1 to 5]
  24 - 48 hours postoperatively | 1 [0 to 4] | 1 [0 to 4]
  48 - 72 hours postoperatively | 2 [0 to 4] | 1 [0 to 3]

ADVERSE EVENTS:
Time Frame: Data collected from day of surgery until removal of epidural, on average epidurals were removed between day 1 and 3. Rare clinical scenarios, epidurals can remain as long as 7 days
Arm/Group | Continuous Epidural Infusion | Programmed Intermittent Epidural Bolus
All-Cause Mortality (participants affected / at risk) | 0/44 | 0/52
Serious Adverse Events (participants affected / at risk) | 0/44 | 0/52
Other Adverse Events (participants affected / at risk) | 9/44 | 18/52
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Continuous Epidural Infusion (N=44) | Programmed Intermittent Epidural Bolus (N=52)
Hypotension (Cardiac disorders) | 9 | 18 — mean arterial blood pressure less than 60

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-07-30): https://cdn.clinicaltrials.gov/large-docs/74/NCT03307174/Prot_SAP_000.pdf